CLINICAL TRIAL: NCT05449639
Title: Multicentric Pilot Study for the Application of a Magnetic Endourethral Sphincter for the Treatment of Secondary Stress Urinary Incontinence Damage to the Urethral Sphincter
Brief Title: Study for a Magnetic Endourethral Sphincter Against Stress Urinary Incontinence
Acronym: RELIEF-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Relief srl (Industry)
Collaborators: Donawa Lifescience (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-002
Record Dates: First submitted 2022-06-07; First posted 2022-07-08 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main group (Experimental): A second no-random open interventional pilot study sponsored by Relief srl. The primary objectives of the study were to assess the safety and reproducibility of the implantation of the magnetic endo-urethral sphincter, if the procedure was well tolerated by the patients, and if possible irritation symptoms due to the device presence emerged in patients with severe stress urinary incontinence where standard medical treatments failed. The device will be implanted by endoscopic procedure by a standard resectoscope. Up to 20 patients of both gender affected by severe stress urinary incontinence will be involved in the study by means of prospective enrollment.
  Interventions: Device: Relief implantation

INTERVENTIONS:
Device: Relief implantation — The device will be implanted by endoscopic procedure by a standard resectoscope.

SUMMARY:
A second no-random open interventional pilot study sponsored by Relief srl

DETAILED DESCRIPTION:
The first pilot study, where the device was implanted on 6 human patients for 28 days, demonstrated that the magnetic urethral sphincter was successfully implanted and explanted in all patients (5 males and 1 female). All the procedures have proven ease of implantation and removal (6/6, 100%), decent simplicity of the activation and de-activation system and restoring an acceptable urinary continence. The majority of patients (5/6, 83.4%) reported a good tolerability of the sphincter. Unfortunately, only 1/6 patient (16.7%) was able to complete the 28 days cycle with the urinary sphincter in place: in the other 5 patients (83.3%) the sphincter migrated into the bladder due to the lack of a hooking system, which was not considered relevant in the design phase and during previous cadaver tests. This migration seemed caused by an oversized external magnet, producing a large force also in not optimized positioning, and by the anatomic variability of patients' urethral caliber. In one patient the sphincter stayed perfectly in place for all the 28 days; its position was checked after 10 days of the implantation by suprapubic ultrasound scan. This patient referred excellent urinary continence also with the sphincter in the "opened" configuration (without using the external magnet but by relying only on the valve flexibility), without urinary leaks during daily activities and sport activities too. No severe side effects or complications or infections occur after the migration of the device in the bladder and during its implantation/removal.

The final analysis of data and questionnaires showed that, to adapt the magnetic urethral sphincter to the clinical practice, a re-design is necessary in order to improve the anchoring system and to optimize the magnetic activation system, avoiding bladder migration of the device.

In this framework Relief re-designed the device by optimizing the external magnet, by improving the proximal anchoring system and by providing with a distal anchoring system. The new design was validated by test bench and on cadaver anatomies.

The primary objectives of the study were to assess the safety and reproducibility of the implantation of the magnetic endo-urethral sphincter, if the procedure was well tolerated by the patients, and if possible irritation symptoms due to the device presence emerged in patients with severe stress urinary incontinence where standard medical treatments failed.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged from 45 to 85 years-old suffering from secondary Stress Urinary Incontinence (SUI) to prostate surgery in which medical and rehabilitative treatment have failed;
2. women patients aged from 45 to 85 years-old suffering from SUI in which medical, rehabilitative and surgical treatment have failed;
3. sterile urine culture;
4. urodynamic test with evidence of sphincter dysfunction, Valsalva Leak Point Pressure (VLPP) < 60 cm H2O (water) and exclusion of detrusor over-activity;
5. flexible cystoscopy demonstrating sphincter dysfunction and excluding stenosis of the urethra or vesicourethral anastomosis.

Exclusion Criteria:

1. No-autonomous patients;
2. People where the use of magnetic field is not suggested (i.e. patients with pacemaker).
3. Patients with urinary infections;
4. Patients with intolerances to the materials included in the sphincter or to expected drug subministration.
5. Patients already participating a clinical study within the last 30 days.
6. Patients that already have devices/solutions or part of them for the treatment of urinary incontinence.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Absence of post-operative symptoms | 90 days
  The primary end-point regarding the tolerability and safety of the device will be verified by interviewing the patient about the appearance of post-operative irritative symptoms and the ease of use of the system. The outcome will be evaluated on the basis of the onset of any surgical complications according to the Clavien-Dindo classification. This classification (consisting of 7 grades such as I, II, IIIa, Illb, IVa, IVb, V) is widely used and has become the standard classification system for many surgical specialties.
Performance of the implantation | 60 days
  Implant performance will be assessed in terms of implant migration via an ultrasound at 10, 30 and 60 days after the application of the magnetic endourethral sphincter, in order to verify the correct positioning and stability of the device.

SECONDARY OUTCOMES:
Efficacy of the implantation on the disease | 90 days
  The secondary end-point about the efficacy of the magnetic endourethral sphincter by the patient will be evaluated through the validated qualitative International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF) administered before starting the procedure, at 10, 30, 60 and 90 days.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Casa di Cura San Camillo, Forte dei Marmi, Lucca
  - Azienda Ospedaliero Universitaria Pisana UO Urologia, Pisa
  - Policlinico Universitario Campus Bio-Medico UOC Urologia, Roma

IPD SHARING:
Plan to Share IPD: No
The results of this study will be presented at appropriate conferences and presented for publication in peer-reviewed journals. The publication will be completed in line with the contract.
  The Study Sponsor will collect the data in such a way that no subjects can be identified and will monitor the study records. Participating subjects will not be identified by name in any published study reports.